CLINICAL TRIAL: NCT00022217
Title: A Phase II Activity And Safety Study Of IntraDose (Cisplatin/Epinephrine Injectable Gel) When Given In Combination With Systematic Chemotherapy Paclitaxel And Carboplatin In The Treatment Of Patients With Squamous Cell Carcinoma Of The Head And Neck At First Relapse
Brief Title: Cisplatin-Epinephrine Injectable Gel Plus Paclitaxel and Carboplatin in Treating Patients With Recurrent Head and Neck Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Matrix Pharmaceutical (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068796; MP-601-00-2; ENH-EH01-102
Record Dates: First submitted 2001-08-10; First posted 2004-02-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2002-02

CONDITIONS: Head and Neck Cancer
Keywords: recurrent salivary gland cancer; salivary gland squamous cell carcinoma; salivary gland anaplastic carcinoma; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent verrucous carcinoma of the oral cavity; recurrent squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Carboplatin; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin-e therapeutic implant
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving more than one drug and giving the drugs in different ways may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of cisplatin-epinephrine injectable gel plus paclitaxel and carboplatin in treating patients who have recurrent head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the antitumor activity of intratumoral cisplatin-epinephrine injectable gel and systemic paclitaxel and carboplatin in patients with recurrent squamous cell carcinoma of the head and neck. II. Determine the safety of this regimen in this patient population. III. Determine the time to progression, pattern of progression, and rate of relapse of patients treated with this regimen. VI. Determine the time to response and duration of response of patients treated with this regimen. V. Determine the overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients receive cisplatin-epinephrine gel intratumorally on days -15, -8, 1, 8, 15, and 22 for course 1 and days 1, 8, 15, and 22 for all subsequent courses. Patients also receive paclitaxel IV over at least 3 hours followed by carboplatin IV over at least 30 minutes on day 1. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients who achieve local complete response (CR) and no metastatic disease progression continue treatment with carboplatin and paclitaxel only. Patients who achieve total CR may receive 2 additional courses of carboplatin and paclitaxel. Patients are followed at 1-4 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: Approximately 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent primary squamous cell carcinoma of the head and neck The following other histological types are also eligible: Epithelial carcinoma Verrucous carcinoma Sarcomatoid squamous cell carcinoma Lymphoepithelioma Pseudosarcoma Anaplastic carcinoma Transitional cell carcinoma At first relapse after prior definitive surgery, radiotherapy, and/or chemotherapy and not a candidate for potentially curative salvage surgery or salvage radiotherapy Relapsed or metastatic disease in one of the following primary head and neck areas or other metastatic sites of skin or soft tissue accessible for local injection: Oral cavity (including tongue, floor of mouth, uvula, and tonsil) Hypopharynx Larynx Nasopharynx Paranasal sinus Salivary gland Tridimensionally measurable disease Tumor no greater than 20 cm3 At no immediate risk of invasion of a major vessel of the extracranial vascular system (e.g., the common, internal, or external carotid artery or the vertebral artery) Amenable to direct injection by physical exam, ultrasound, or CT guidance Visceral metastases (e.g., lung) allowed but not eligible for injection with cisplatin-epinephrine gel

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Platelet count at least 100,000/mm3 Neutrophil count at least 1,500/mm3 Hemoglobin at least 10 g/dL Hepatic: Bilirubin less than 3 mg/dL AST no greater than 3 times upper limit of normal (ULN) Alkaline phosphatase no greater than 3 times ULN Albumin no greater than 2.5 g/dL PT within 3 seconds of normal Renal: Creatinine no greater than 1.5 times ULN OR Creatinine clearance at least 50 mL/min Cardiovascular: See Disease Characteristics No New York Heart Association class III or IV heart disease Other: No other malignancy within the past 5 years except nonmelanoma skin cancer outside the area of planned cisplatin-epinephrine gel treatment No known hypersensitivity to cisplatin, carboplatin, paclitaxel, bovine collagen, epinephrine, or sulfites No infection requiring parenteral antibiotics No medical or psychiatric condition that would preclude informed consent Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 28 days since prior chemotherapy and recovered Prior carboplatin or taxanes allowed, but not in combination Endocrine therapy: Concurrent stable-dose prednisone/prednisolone for chronic disease allowed Concurrent stable-dose corticosteroid inhalants for asthma prophylaxis allowed Concurrent dexamethasone as an antiemetic allowed Radiotherapy: See Disease Characteristics At least 28 days since prior radiotherapy and recovered Concurrent limited-field radiotherapy for symptomatic metastatic disease not amenable to cisplatin-epinephrine gel allowed Surgery: See Disease Characteristics At least 28 days since prior surgery and recovered Other: No concurrent anesthetics or topical preparations containing epinephrine No other concurrent cancer therapy No drugs that interact with cisplatin (e.g., probenecid or thiazide) during and for 28 days after study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-11

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Elias, MD, Study Chair — Matrix Pharmaceutical
Locations (4):
- United States (4):
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Division of Head and Neck Surgery, Evanston, Illinois
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana